CLINICAL TRIAL: NCT00372697
Title: A Randomised, Open-label, Multicenter Study Comparing the Efficacy and Safety of Medical Treatment With Octreotide Acetate 30 mg Administered Every 21 Days for 6 Months With That of Octreotide Acetate 60 mg Administered Every 28 Days for 6 Months in Acromegalic Patients With Uncontrolled Disease
Brief Title: Efficacy/Safety of Octreotide Acetate in Patients With Uncontrolled Acromegaly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSMS995BIT12
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Results first posted 2011-05-17 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-04

CONDITIONS: Acromegaly
Keywords: acromegaly; octreotide acetate; partial responder patients
MeSH Terms: conditions — Acromegaly | interventions — Octreotide; Suspensions

ARMS (2):
- Octreotide 30 mg every 21 days (Experimental): Patients received octreotide 30 mg every 21 days intramuscularly (im) for 6 months, a total of 8 doses. At each study visit, octreotide was administered only after completion of all scheduled efficacy and safety evaluations for that visit. Octreotide was injected im into the right or left gluteal regions. The injections were initially administered by a trained and authorized member of the investigational team. When no study visit at the investigational site was required, the injections were given by a trained nurse or the family doctor.
  Interventions: Drug: Octreotide acetate 30 mg suspension
- Octreotide 60 mg every 28 days (Experimental): Patients received octreotide 60 mg every 28 days intramuscularly (im) for 6 months, a total of 6 doses. Octreotide mg was administered as two 30 mg injections. At each study visit, octreotide was administered only after completion of all scheduled efficacy and safety evaluations for that visit. Octreotide was injected im into the right or left gluteal regions. The injections were initially administered by a trained and authorized member of the investigational team. When no study visit at the investigational site was required, the injections were given by a trained nurse or the family doctor.
  Interventions: Drug: Octreotide acetate 30 mg suspension

INTERVENTIONS:
Drug: Octreotide acetate 30 mg suspension — Each vial of study medication contained octreotide acetate 30 mg in a microencapsulated biodegradable polymer, poly (DL-lactide-co-glycolide) (D-(+)glucose), with 17% w/w mannitol in an approximate octreotide:polymer ratio of 1:20. The vehicle contained 0.5% sodium carboxymethylcellulose.
  Other Names: Sandostatin LAR

SUMMARY:
This study evaluated the safety and efficacy of an increased frequency of octreotide acetate injections or an increase in dose in partially responsive acromegalic patients with persistently uncontrolled disease.

ELIGIBILITY:
Inclusion Criteria:

* Written voluntary informed consent.
* Patients with biochemically documented active acromegaly who are currently receiving somatostatin-analogues in a conventional treatment regimen (octreotide up to 30 mg/28 days; lanreotide up to 120 mg/28 days) for at least 6 months.
* Patients with uncontrolled disease defined as patients with a decrease of baseline levels of growth hormone (GH) ≥ 50% during treatment with somatostatin-analogues in a conventional regimen (sandostatin up to 30 mg/28 days; lanreotide up to 120 mg/28 days) for at least 6 months.
* Baseline (mean of 3 samples) GH level > 2 µg/L.
* Insulin-like Growth Factor I (IGF-I) levels above the upper limits of normal for age and gender.

Other protocol-defined inclusion/exclusion criteria applied to the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- Novartis Investigative Site, Brescia, Italy

REFERENCES:
- [Derived] Mazziotti G, Porcelli T, Bogazzi F, Bugari G, Cannavo S, Colao A, Cozzi R, De Marinis L, degli Uberti E, Grottoli S, Minuto F, Montini M, Spinello M, Giustina A. Effects of high-dose octreotide LAR on glucose metabolism in patients with acromegaly inadequately controlled by conventional somatostatin analog therapy. Eur J Endocrinol. 2011 Mar;164(3):341-7. doi: 10.1530/EJE-10-0811. Epub 2011 Jan 6. PMID 21212103

RESULTS

PARTICIPANT FLOW:
Groups:
- Octreotide 30 mg Every 21 Days: Participants received octreotide 30 mg every 21 days intramuscularly (im) for 6 months, a total of 8 doses. At each study visit, octreotide was administered only after completion of all scheduled efficacy and safety evaluations for that visit. Octreotide was injected im into the right or left gluteal regions. The injections were initially administered by a trained and authorized member of the investigational team. When no study visit at the investigational site was required, the injections were given by a trained nurse or the family doctor.
- Octreotide 60 mg Every 28 Days: Participants received octreotide 60 mg every 28 days intramuscularly (im) for 6 months, a total of 6 doses. Octreotide mg was administered as two 30 mg injections. At each study visit, octreotide was administered only after completion of all scheduled efficacy and safety evaluations for that visit. Octreotide was injected im into the right or left gluteal regions. The injections were initially administered by a trained and authorized member of the investigational team. When no study visit at the investigational site was required, the injections were given by a trained nurse or the family doctor.
Period: Overall Study
Arm/Group | Octreotide 30 mg Every 21 Days | Octreotide 60 mg Every 28 Days
Started | 16 | 12
Completed | 15 | 11
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Octreotide 30 mg Every 21 Days | Octreotide 60 mg Every 28 Days | Total
Number analyzed (Participants) | 16 | 12 | 28
Age Continuous [Mean (Standard Deviation); unit: years] | 51.3 (12.1) | 51.8 (15.7) | 51.5 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14
  Male | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Growth Hormone (GH) Level From Screening to End of Study (Week 24)
Description: Growth hormone (GH) level was the average value measured in 3 blood samples collected at 15 minute intervals at each visit. GH was measured with an automated immunometric assay in a central laboratory.
Time Frame: Screening to end of study (Week 24)
Population: Intent-to-treat (ITT) population included all participants who received at least one dose of study medication and who had at least one post-baseline evaluation of the primary variable.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Octreotide 30 mg Every 21 Days | Octreotide 60 mg Every 28 Days
Number analyzed (Participants) | 15 | 11
µg/L | -1.7 (9.9) | -2.1 (3.6)

2. Primary Outcome: Change in Insulin-like Growth Factor 1 (IGF-1) Level From Screening to End of Study (Week 24)
Description: Insulin-like growth factor 1 (IGF-1) level was measured in a blood sample with an automated immunometric assay in a central laboratory.
Time Frame: Screening to end of study (Week 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Octreotide 30 mg Every 21 Days | Octreotide 60 mg Every 28 Days
Number analyzed (Participants) | 15 | 11
µg/L | -40.4 (180.2) | -135.0 (170.9)

3. Secondary Outcome: Change in Tumor Volume From Screening to End of Study (Week 24)
Description: A pre-treatment magnetic resonance image (MRI) assessment of the pituitary area was required within 12 weeks prior to Screening as a baseline evaluation. A second MRI was performed at the end of the study (Week 24). All MRIs were performed according to protocol-defined guidelines. The tumor volume (mm^3) was calculated from measurements obtained in 3 axes from the MRI images.
Time Frame: Screening to end of study (Week 24)
Population: Intent-to-treat (ITT) population included all enrolled participants who received at least 1 dose of assigned study medication and who had data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Octreotide 30 mg Every 21 Days | Octreotide 60 mg Every 28 Days
Number analyzed (Participants) | 14 | 9
mm^3 | 15.9 (91.8) | -0.4 (21.0)

4. Secondary Outcome: Percentage of Participants With > 20% Tumor Shrinkage From Screening to End of Study (Week 24)
Description: as for outcome 3
Time Frame: Screening to end of study (Week 24)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Octreotide 30 mg Every 21 Days | Octreotide 60 mg Every 28 Days
Number analyzed (Participants) | 14 | 9
Percentage of participants | 14.3 (6426) | 11.1 (4211)

5. Secondary Outcome: Percentage of Participants Asymptomatic for Acromegaly Symptoms at Week 12 and End of Study (Week 24)
Description: The investigator asked the participant to score the following symptoms of acromegaly: Headache, perspiration, paresthesia, fatigue, osteoarthralgia, and carpal tunnel syndrome on a 5-point scale (0=absent; 1=mild; 2=moderate; 3=severe, but not disabling; 4=severe and disabling). The percentage of asymptomatic participants, ie, with a score of 0 for all symptoms, was calculated.
Time Frame: Week 12 and end of study (Week 24)
Population: Intent-to-treat (ITT) population included all enrolled participants who received at least 1 dose of assigned study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Octreotide 30 mg Every 21 Days | Octreotide 60 mg Every 28 Days
Number analyzed (Participants) | 15 | 11
Percentage of participants
  Week 12 | 33.3 | 9.09
  Week 24 | 20.0 | 9.09

6. Secondary Outcome: Acromegaly Quality of Life (AcroQoL) Questionnaire Physical Scale Score at End of Study (Week 24)
Description: The AcroQoL contains 8 items on Physical aspects. Participants were asked to rate each item on a 1-5 Likert scale measuring either the frequency of occurrence (always, most of the time, sometimes, rarely, or never) or the degree of agreement (completely agree, moderately agree, neither agree nor disagree, moderately disagree, completely disagree). The score on the physical scale can range from 8-40. A higher score indicates better Quality of Life.
Time Frame: End of study (Week 24)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent of maximum score
Arm/Group | Octreotide 30 mg Every 21 Days | Octreotide 60 mg Every 28 Days
Number analyzed (Participants) | 15 | 11
Percent of maximum score | 67.9 (22.6) | 58.0 (21.8)

7. Secondary Outcome: Acromegaly Quality of Life (AcroQoL) Questionnaire Psychological Scale Score at End of Study (Week 24)
Description: The AcroQoL contains 14 items on Psychological aspects. Participants were asked to rate each item on a 1-5 Likert scale measuring either the frequency of occurrence (always, most of the time, sometimes, rarely, or never) or the degree of agreement (completely agree, moderately agree, neither agree nor disagree, moderately disagree, completely disagree). The score on the psychological scale ranges from 14-70. A higher score indicates better Quality of Life.
Time Frame: End of study (Week 24)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent of maximum score
Arm/Group | Octreotide 30 mg Every 21 Days | Octreotide 60 mg Every 28 Days
Number analyzed (Participants) | 15 | 10
Percent of maximum score | 65.1 (19.9) | 72.1 (19.6)

ADVERSE EVENTS:
Arm/Group | Octreotide 30 mg Every 21 Days | Octreotide 60 mg Every 28 Days
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 3/16 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octreotide 30 mg Every 21 Days (N=16) | Octreotide 60 mg Every 28 Days (N=12)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.